CLINICAL TRIAL: NCT04253964
Title: Phase II Pilot Study of Performance Status 2 vs. Performance Status 0-1 Non-Small Cell Lung Cancer Patients Treated With Chemo/Immunotherapy
Brief Title: Pilot Study of Performance Status 2 vs. Performance Status 0-1 Non-small Cell Lung Cancer Patients Treated With Chemo/Immunotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00063540; WFBCCC 62619 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Nonsmall Cell Lung Cancer; Performance Status
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Carboplatin; Paclitaxel; Taxes; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Performance Status 0-1 Participants (Experimental): ALL study participants will receive pembrolizumab 200 mg intravenously (IV) on day 1 of each 3-week cycle.
  Participants with predictive biomarker PD-L1 greater than or equal to 50%: Participants will not receive any other drugs besides pembrolizumab.
  Participants with Non-squamous subtype, predictive biomarker (PD-L1 less than 50%): Participants will ALSO receive:
  - Carboplatin area under the curve (AUC) 5 IV on day 1 of each 3-week cycle for 4 cycles.
  PLUS
  - Pemetrexed 500 mg/m2 IV on day 1 of each 3-week cycle for 4 cycles.
  Participants with Squamous subtype, predictive biomarker (PD-L1 less than 50%): Participants will also receive:
  * Carboplatin AUC 5 IV on day 1 of each 3-week cycle for 4 cycles. PLUS
  * Paclitaxel 200 mg/m2 IV on day 1 of each 3-week cycle for 4 cycles. OR
  * Nab-paclitaxel 100 mg/m2 on day 1, 8, 15 of 3-week cycle for 4 cycles
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab paclitaxel; Other: Quality of Life Questionnaire, lung cancer-specific (QLQ-LC13); Other: QLQ-C30 Global Health/Quality of Life Questionnaire; Other: COPD Assessment Test and modified Medical Research Council Dyspnea Patient Reported Outcomes; Drug: Pemetrexed
- Performance Status 2 Participants (Experimental): ALL study participants will receive pembrolizumab 200 mg intravenously (IV) on day 1 of each 3-week cycle.
  Participants with predictive biomarker PD-L1 greater than or equal to 50%: Participants will not receive any other drugs besides pembrolizumab.
  Participants with Non-squamous subtype, predictive biomarker (PD-L1 less than 50%): Participants will ALSO receive:
  - Carboplatin area under the curve (AUC) 5 IV on day 1 of each 3-week cycle for 4 cycles.
  PLUS
  - Pemetrexed 500 mg/m2 IV on day 1 of each 3-week cycle for 4 cycles.
  Participants with Squamous subtype, predictive biomarker (PD-L1 less than 50%): Participants will also receive:
  * Carboplatin AUC 5 IV on day 1 of each 3-week cycle for 4 cycles. PLUS
  * Paclitaxel 200 mg/m2 IV on day 1 of each 3-week cycle for 4 cycles. OR
  * Nab-paclitaxel 100 mg/m2 on day 1, 8, 15 of 3-week cycle for 4 cycles
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab paclitaxel; Other: Quality of Life Questionnaire, lung cancer-specific (QLQ-LC13); Other: QLQ-C30 Global Health/Quality of Life Questionnaire; Other: COPD Assessment Test and modified Medical Research Council Dyspnea Patient Reported Outcomes; Drug: Pemetrexed

INTERVENTIONS:
Drug: Pembrolizumab — ALL PARTICIPANTS: Pembrolizumab 200 mg intravenously (IV) on day 1 of each 3-week cycle for 4 cycles. Participants with predictive biomarker PD-L1 greater than or equal to 50% will not receive any other drugs besides pembrolizumab.
Drug: Carboplatin — FOR PARTICIPANTS IN EITHER ARM with non-squamous OR squamous subtype, predictive biomarker PD-L1 less than 50%: Carboplatin area under the curve (AUC) 5 IV on day 1 of each 3-week cycle for 4 cycles.
Drug: Paclitaxel — FOR PARTICIPANTS IN EITHER ARM with squamous subtype, predictive biomarker PD-L1 less than 50%: Paclitaxel 200 mg/m2 IV on day 1 of each 3-week cycle for 4 cycles.
Drug: Nab paclitaxel — FOR PARTICIPANTS IN EITHER ARM with squamous subtype, predictive biomarker PD-L1 less than 50%: Nab-paclitaxel 100 mg/m2 on day 1, 8, 15 of 3-week cycle for 4 cycles.
Other: Quality of Life Questionnaire, lung cancer-specific (QLQ-LC13) — The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
Other: QLQ-C30 Global Health/Quality of Life Questionnaire — 30 item questionnaire - Functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, and nausea and vomiting), global health status and quality of life scale, also several single-item symptom measures
Other: COPD Assessment Test and modified Medical Research Council Dyspnea Patient Reported Outcomes — Dyspnea scale scores in patients with respiratory disease (particularly COPD) to establish baseline functional dyspnea burden (taken pre-study at Week 0 and Post Treatment at week 13)
Drug: Pemetrexed — FOR PARTICIPANTS IN EITHER ARM with nonsquamous subtype, predictive biomarker PD-L1 less than 50%: Pemetrexed 500 mg/m2 IV on day 1 of each 3-week cycle for 4 cycles.

SUMMARY:
This pilot study is configured as a non-inferiority comparison of Performance Status 2 patients with Performance Status 0-1 patients, with the goal of demonstrating non-inferiority in terms of efficacy (progression-free survival, overall survival) and safety (rates of adverse events, quality of life) when treating Performance Status 2 patients with the same first-line immunotherapy-based regimen as Performance Status 0-1 patients.

DETAILED DESCRIPTION:
Primary Objective: To demonstrate that proportion of Performance Status 2 participants with progression-free survival at 12 weeks is not inferior to the corresponding proportion of Performance Status 0-1 patients.

Secondary Objective(s)

* To demonstrate that incidence of treatment-related adverse events at 12 weeks in the Performance Status 2 group is not higher than that occurring in the Performance Status 0-1 groups.
* To demonstrate that change in overall quality of life/global health status at 12 weeks is not inferior in the Performance Status 2 group compared to the change in the Performance Status 0-1 group.
* To demonstrate that proportion of participants with deterioration in lung-cancer specific symptoms at 12 weeks in the Performance Status 2 group is not higher than the corresponding proportion in the Performance Status 0-1 group.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a cytological or histological diagnosis of non-small cell lung cancer that is metastatic or unresectable for which standard curative measures do not exist.
* No prior systemic treatment with either chemotherapy or immunotherapy for non-curative intent. Patients may have previously received cancer treatment with curative intent for prior early-stage disease.
* At least 18 years old.
* ECOG performance status of 0-2, as determined by the treating physician in the consult note.
* Life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function as defined below:
* absolute neutrophil count ≥1,000/mcL
* platelets ≥100,000/mcL
* Chemotherapy agents are known to be teratogenic, therefore women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign an IRB-approved informed consent document.

Exclusion Criteria:

* Nonsmall cell lung cancer that is known at registration to be positive for a tumor activating alteration for which first line targeted therapy is indicated; specifically, a targetable mutation in epidermal growth factor receptor (EGFR), gene rearrangement of anaplastic lymphoma kinase (ALK), gene rearrangement of c-ros oncogene 1 (ROS1), or mutation in B isoform of rapidly accelerated fibrosarcoma (B-Raf). For non-squamous subtypes, molecular testing of tumor and peripheral blood should be attempted for actionable biomarkers, but if there is an insufficient quantity of tumor material for testing and it is not feasible to attempt additional biopsies before starting systemic therapy, then these biomarker results are not necessary for inclusion on the study. For squamous subtype, molecular testing should be considered but is not necessary for inclusion on the study.
* Known to have an active autoimmune disease that required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, systemic corticosteroids, or immunosuppressive drugs).
* History of (non-infectious) pneumonitis that required systemic corticosteroids.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects with chemotherapy. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with chemotherapy, breastfeeding should be discontinued.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with Progression-Free Survival | From baseline to end of 4th cycle of treatment (12 weeks)
  Using non-blinded central imaging using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 to define progressive disease.
  RECIST v 1.1 criteria:
  * Complete Response (CR): Disappearance of all target lesions.
  * Partial Response (PR): Decrease by ≥ 30% in sum of longest diameter of target lesions.
  * Stable Disease (SD): Not meeting criteria for CR, PR, or PD.
  * Progressive Disease (PD): Increase by ≥ 20% in sum of longest diameter of target lesions or the appearance of one or more new lesions.
  Participants that did not have radiographically measurable metastatic disease by RECIST criteria before starting treatment, progression is defined as the development of new lesions or by unequivocal progression of existing non-target lesions.

SECONDARY OUTCOMES:
Incidences of Grade 3 to Grade 5 Treatment-Related Adverse Events | 12 weeks
  Adverse events will be defined using CTCAE Version 5.0 after four cycles (12 weeks).
Change in Overall Quality of Life/Global Health Status - EORTC QLQ-C30 | From baseline to end of 4th cycle of treatment (12 weeks)
  Using the total score of the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30), a 30-item questionnaire for functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, and nausea and vomiting), global health status and quality of life scale, also several single-item symptom measures. Scoring scale : 1 (Not at all) to 4 (Very much), 1 (Very poor) to 7 (Excellent). Minimum score 0, maximum score 100. For functional and global quality of life scales, higher scores mean a better level of functioning. For symptom-oriented scales, a higher score means more severe symptoms.
Proportion of Participants with Deterioration in Symptoms - QLQ-LC13 | From baseline to end of 4th cycle of treatment (12 weeks)
  Patient reported deterioration in three symptoms: Cough, chest pain, or dyspnea as measured by the symptoms scales as part of the Quality of Life Questionnaire Lung Cancer Module (QLQ-LC13). Deterioration is defined as a 10-point or greater decrease from baseline in either cough, chest pain, or dyspnea and subsequently confirmed by a second adjacent 10-point or greater decrease from baseline in the same symptom)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lycan, Jr., D.O., M.H.S., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No